CLINICAL TRIAL: NCT06462300
Title: Searching for Meaning: A Study Examining the Effect of a Meaning-centered Intervention
Brief Title: Meaning-centered Intervention for Young Women With Weight and Shape Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSY-2223-S-0010
Record Dates: First submitted 2024-06-03; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Eating Disorder Symptom
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning-centered intervention condition (Experimental): The group of participants receiving the meaning-centered intervention
  Interventions: Behavioral: A meaning-centered intervention for young women with weight and shape concerns
- Waitlist control condition (No Intervention): The group of participants not receiving an intervention

INTERVENTIONS:
Behavioral: A meaning-centered intervention for young women with weight and shape concerns — * adapted version of the manualized meaning-centered psychotherapy for cancer patients developed by van der Spek et al. (2017)
  * six weekly individual online sessions, each lasting one hour
  * sessions led by a certified trainer
  * four sources of meaning will be explored: personal life story, dealing with life's limitations, creating one's own life, and meaningful experiences
  * homework assignments designed to deepen participants' experience and reflection on meaning in their daily lives
  Arms: Meaning-centered intervention condition

SUMMARY:
Female participants with weight and shape concerns will either receive a six-week meaning-centered intervention led by a trainer or be allocated to a waitlist condition. They will receive the same questionnaires at three time points: Before the intervention, immediately after, and four weeks later.

The researchers hypothesize that a meaning-centered intervention for young women with weight and shape issues will increase participants meaning in life and decrease their eating disorder symptoms immediately after the intervention and at 4-week follow-up when compared to a waitlist condition.

DETAILED DESCRIPTION:
Female first-year psychology students at the University of Groningen will be screened for weight and shape concerns. Those scoring in the clinically relevant range will be invited to participate in the study. After filling out the baseline measures online, the participants will be randomly allocated to a waitlist or an intervention condition. Participants in the intervention condition will follow a weekly 1-hour online intervention with a trainer for six weeks, including homework assignments. In this intervention, the aim is to increase meaning in life and decrease eating disorder symptoms. All study materials will be offered in English, Dutch, or German. Immediately after the intervention and four weeks later, the participants will receive the same questionnaires again as at baseline. The waitlist participants will not receive any intervention during the six-week period between baseline and post-assessment, but receive the same questionnaires in the same timeframe. Waitlist participants will also have the option to receive the intervention after the study has been finished.

ELIGIBILITY:
Inclusion Criteria:

* When screened with the Weight Concerns Scale (WCS; Killen et al., 1994) and when scores of all five items were adjusted to equal a maximum score of 20, leading to a total range between 0 and 100 (cf. Jacobi et al., 2004), participant are eligible if they answer "always" or "often" to the item "Do you ever feel fat?" or have a total score ≥ 47 on the WCS or both

Exclusion Criteria:

* Current treatment for eating disorder
* not fluent in English, Dutch, or German

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants had to indicate "woman" as their preferred gender identity during the screening process.
Enrollment: 166 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Meaning in life | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Presence of meaning in life subscale of Meaning in Life Questionnaire (Steger et al., 2006); average of 5 items with 7-point Likert scale (minimum: 1; maximum 7); the higher the score, the higher the presence of life meaning

SECONDARY OUTCOMES:
Tripartite domain of meaning in life: Comprehension | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Comprehension subscale of Multidimensional Existential Meaning Measure (George & Park, 2016); average of 5 items on 7-point Likert scale (minimum: 1; maximum: 7); the higher the score, the higher the sense of Comprehension
Tripartite domain of meaning in life: Purpose | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Purpose subscale of Multidimensional Existential Meaning Measure (George & Park, 2016); average of 5 items on 7-point Likert scale (minimum: 1; maximum: 7); the higher the score, the higher the sense of Purpose
Tripartite domain of meaning in life: Mattering | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Mattering subscale of Multidimensional Existential Meaning Measure (George & Park, 2016); average of 5 items on 7-point Likert scale (minimum: 1; maximum: 7); the higher the score, the higher the sense of Mattering
Eating disorder symptoms | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Global score of Eating Disorder Examination-Questionnaire (Fairburn & Beglin, 2008); average score of 22 items on a 7-point Likert scale (minimum: 0; maximum: 6); the higher the score, the more severe the eating disorder symptomatology
Internalizing symptoms | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Total score of Depression Anxiety Stress Scales-21 (Lovibond & Lovibond, 1995); sum score of 21 items on a 4-point Likert scale (minimum: 0; maximum: 63); the higher the score, the more severe the internalizing symptomatology
Depressive symptoms | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Depression subscale of Depression Anxiety Stress Scales-21 (Lovibond & Lovibond, 1995); sum score of 7 items on a 4-point Likert scale (minimum: 0; maximum: 21); the higher the score, the more severe the depressive symptomatology
Anxiety symptoms | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Anxiety subscale of Depression Anxiety Stress Scales-21 (Lovibond & Lovibond, 1995); sum score of 7 items on a 4-point Likert scale (minimum: 0; maximum: 21); the higher the score, the more severe the anxiety symptoms
Stress symptoms | Baseline (week 1), post-assessment (week 7), follow-up (week 11)
  Stress subscale of Depression Anxiety Stress Scales-21 (Lovibond & Lovibond, 1995); sum score of 7 items on a 4-point Likert scale (minimum: 0; maximum: 21); the higher the score, the more severe the stress symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies the results in the finalized publication will be made available
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Access will be given based on individual requests

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT06462300/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT06462300/ICF_001.pdf